CLINICAL TRIAL: NCT04232501
Title: Effect of Novel Sequential Compression Device on the Incidence of Deep Venous Thrombosis on Complex Surgical Spine Patients
Brief Title: Radial, Sequential Compression Device Deep Venous Thrombosis Detection Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, Radial slowed their operations. Hence the investigational device is not available.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Adam Schlifke, Clinical Assistant Professor, Anesthesia, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-54247
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cirvo Compression device post surgery (Experimental): Patients will wear Cirvo compression device during the surgery, after surgery and will be discharged to home with the device to wear at home as the per study protocol instructions.
  Interventions: Device: Cirvo Compression device
- Standard of Care Post Surgery (No Intervention): Patients receive standard-issue SCDs (pneumatic compression) and wear in surgery and after surgery until they are discharged home.

INTERVENTIONS:
Device: Cirvo Compression device — Patients will wear Cirvo compression device during the surgery, after surgery and will be discharged to home with the device to wear at home as the per study protocol instructions.
  Arms: Cirvo Compression device post surgery

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new leg compression device in preventing post-surgical deep vein thrombosis (blood clot) that can occur after major and complex spine surgery. The investigators aim to show that this new compression device is no worse than the standard sequential compression device (SCD) at preventing DVT and may be able to detect deep vein thrombosis in patients who are not typically screened for this diagnosis after surgery. This new device may be able to capture an important post-surgical complication while providing a more comfortable treatment option.

DETAILED DESCRIPTION:
Compression therapy of the leg is a proven and well-established modality to prevent deep vein thrombosis in immobilized and post-surgical patients. The investigators aim to compare a new sequential compression for the leg that utilizes a servo motor for compression as opposed to a traditional pneumatic motor that is typically used in the hospital and after surgery. Pneumatic sequential compression devices are cumbersome, expensive and not mobile. This new compression device was developed to provide a cheaper, mobile device that can be worn by the patient after surgery and while at home during ambulation. The addition of the servo motor and fine sensors may also be able to detect sub-clinical DVT's that contribute to post-surgical pulmonary embolus and post-surgical complications. The investigators aim to learn how this new device performs in the subset of patients undergoing complex spine surgery, the incidence of post-surgical DVT with this new device compared to traditional SCD and if this new device is capable of detecting sub-clinical post-surgical DVT.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for complex spine surgery at Stanford Hospital

Exclusion Criteria:

* Pregnancy
* Non-decisional capacity
* Incarcerated persons
* Any hereditary or acquired coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-01-08 (Estimated); Study Completion 2021-01-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Deep Vein Thrombosis (DVT) | Within four weeks after surgery
  Number of participants with DVT diagnosed by ultrasound after complex spine surgery

CONTACTS AND LOCATIONS:
Overall Officials: Adam Schlifke, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No